CLINICAL TRIAL: NCT06680167
Title: A Comparative Study Between Hyperbaric Prilocaine 2% Versus Hyperbaric Bupivacaine 0.5% For Intrathecal Anesthesia in Caesarean Section
Brief Title: Hyperbaric Prilocaine 2% vs Hyperbaric Bupivacaine 0.5% in Caesarean Section
Status: Active, not recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Mostafa Mohamed Abdelgaber, A Comparative Study between Hyperbaric Prilocaine 2% versus Hyperbaric Bupivacaine 0.5% For Intrathecal Anesthesia in Caesarean Section, Sohag University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: Soh-Med-15-10---6MS
Record Dates: First submitted 2024-11-05; First posted 2024-11-08 (Actual); Last update posted 2024-11-08 (Actual); Status verified 2024-11

CONDITIONS: Spinal Anesthesia
Keywords: onset time and duration of action; effects on maternal hemodynamics intraoperative and postoperative; evaluation of pain scores postoperatively
MeSH Terms: interventions — Anesthesia, Spinal

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- patients of group A will receive 60mg of hyperbaric prilocaine 2% for spinal anesthesia (Active Comparator)
  Interventions: Drug: spinal anesthesia (hyperbaric Prilocaine 2%)
- patients of group B will receive 12.5mg heavy bupivacaine for spinal anesthesia (Active Comparator)
  Interventions: Drug: Spinal anesthesia (heavy bupivacaine 0.5%)

INTERVENTIONS:
Drug: Spinal anesthesia (heavy bupivacaine 0.5%) — 12.5mg of Heavy bupivacaine 0.5% will be injected intrathecally for women undergoing elective caesarean section
  Arms: patients of group B will receive 12.5mg heavy bupivacaine for spinal anesthesia
Drug: spinal anesthesia (hyperbaric Prilocaine 2%) — 60mg of Hyperbaric Prilocaine 2% will be injected intrathecally for women undergoing elective caesarean section
  Arms: patients of group A will receive 60mg of hyperbaric prilocaine 2% for spinal anesthesia

SUMMARY:
Comparison between effects of hyperbaric bupivacaine 0.5% vs Hyperbaric prilocaine 2% in spinal anesthesia of women undergoing elective caesarean section such as onset time of sensory and motor block, duration of sensory and motor block, effects of maternal hemodynamics and expected side effects .

DETAILED DESCRIPTION:
Patients will be randomly allocated into two groups:

1. Prilocaine Group (Group A):

   * Patients will receive 60 mg of hyperbaric prilocaine 2% intrathecally.
   * The anesthetic solution will be injected intrathecally using a 25 Gauge spinal needle, with the patient in a sitting position (midline or paramedian technique).
   * The injection will be performed at the L3-L4 or L4-L5 interspace.
2. Bupivacaine Group (Group B):

   * Patients will receive 12.5 mg of hyperbaric bupivacaine 0.5% intrathecally.
   * The anesthetic solution will be injected intrathecally using a 25 Gauge spinal needle, with the patient in a sitting position (midline or paramedian technique) .
   * The injection will be performed at the L3-L4 or L4-L5 interspace.

Procedure Details:

Prior to the procedure, patients will be preloaded with 500 ml of balanced crystalloid solution intravenously. Patients will be positioned in the sitting position for the spinal injection.

The chosen interspace (L3-L4 or L4-L5) will be identified, and the skin will be prepared with an antiseptic solution. A 25 Gauge spinal needle will be used for the intrathecal injection (midline or paramedian technique). After confirming free flow of cerebrospinal fluid, the prepared anesthetic solution will be injected over 10-15 seconds. Following the injection, patients will be placed supine with a slight left lateral tilt to avoid aortocaval compression. The sensory block level will be assessed using Pinprick sensation test, and the motor block will be evaluated using the modified Bromage scale. 5 Blood pressure and heart rate will be monitored every 5 mins until the end of the surgery. In case of hypotension (systolic BP < 90 mmHg or diastolic BP < 60 mmHg), intravenous boluses of 10 mg ephedrine will be administered until blood pressure stabilizes. In case of Bradycardia with Heart rate <55 bpm atropine sulphate 0.01 mg/kg will be given intravenous. Pain Assessment will be done postoperatively via Visual analogue score (VAS) as following if score 3 or less no analgesia required if score 4-5, 1g paracetamol iv will be given if score 6-7, 30mg ketorolac iv will be given if score 7 or more, 2.5mg morphine sulphate iv will be given

ELIGIBILITY:
Inclusion Criteria:

1. Women aged 18-45 years.
2. Patients with uncomplicated pregnancies.
3. American society of anesthesiologist (ASA) physical status I or II.
4. Height between 155 cm and 175 cm.
5. Written informed consent provided. -

Exclusion Criteria:

1. Patients with known allergies to local anesthetics.
2. Contraindications to intrathecal anesthesia (e.g., infection at the injection site and coagulopathy).
3. Severe preeclampsia or eclampsia.
4. Presence of significant comorbidities (e.g., uncontrolled diabetes, hypertension, renal or hepatic dysfunction).
5. History of spinal surgery or significant spinal deformity.
6. Patients who refuse to participate in the study -

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 142 (Estimated)
Dates: Start 2024-10-09 (Actual); Primary Completion 2025-11-05 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Measurment of onset time and duration of sensory block of Hyperbaric Bupivacaine 0.5% and Hyperbaric Prilocaine 2% using pinprick sensation test in women undergoing caesarean section | 12 HOURS
2- Measurment of onset time and duration of motor block of Hyperbaric Bupivacaine 0.5% and Hyperbaric Prilocaine 2% using modified bromage scale in women undergoing caesarean section | 12 hours

CONTACTS AND LOCATIONS:
Locations (1):
- Sohag University Hospitals, Sohag, Sohag Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No
for risk of participant data identification and for privacy concerns